CLINICAL TRIAL: NCT04738760
Title: Clinical Outcomes of High Dose Vitamin D Versus Standard Dose in COVID-19 Egyptian Patients
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Collaborators: Misr International University (Other)
Responsible Party: Principal Investigator, Neven Sarhan, Lecturer at Faculty of Pharmacy, Misr International University
Other Study IDs: COVID-VIT-D
Record Dates: First submitted 2021-02-01; First posted 2021-02-04 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Covid19; Corona Virus Infection; Cytokine Storm; Vitamin D Deficiency
Keywords: COVID-19; Cytokine Storm; Vitamin D
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Cytokine Release Syndrome; Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1: Moderate and severe patients who were infected with SARS-CoV-2 and who were already receiving treatment with standard dose vitamin D in addition to standard COVID-19 management.
- Group 2: Moderate and severe patients who were infected with SARS-CoV-2 and who were already receiving treatment with high dose vitamin Din addition to standard COVID-19 management.

SUMMARY:
Vitamin D is a secosteroid hormone which may have beneficial role in reducing COVID-19 adverse outcomes by first regulating the renin angiotensin system (RAS). Recent studies on animal in which acute respiratory distress syndrome (ARDS) was induced, showed that vitamin D lead to pulmonary permeability reduction by modulating RAS activity as well as the expression of the angiotensin-2 converting enzyme (ACE2). During COVID-19, downregulation of ACE2 leads to cytokine storm in the host, causing ARDS. In contrast, an experimental study conducted on mice in which ARDS was induced chemically, revealed that vitamin D admiration contributed to mRNA and ACE2 proteins levels improvement, ADRS milder symptoms as well as less lung damage.

Additionally, vitamin D had shown antiviral effects on several previous studies, that though to be exerted either by antimicrobial peptides induction which subsequently had direct antiviral action or through immunomodulatory and anti-inflammatory effects.

In addition, vitamin D stabilizes physical barriers which prevent viruses from reaching tissues susceptible to infection. Finally, previous studies demonstrated that hypovitaminosis D is accompanied by various comorbidities including diabetes mellitus, hypertension, chronic cardiovascular and respiratory diseases, and cancers, all medical conditions that are considered risk factors of COVID-19 infection deterioration and even high mortality rate.

The objective of this study is to evaluate whether supplementation with high-dose vitamin D improves the prognosis of patients diagnosed with COVID-19 compared to a standard dose of vitamin D.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 65 years.
2. COVID-19 hospitalized patients with pneumonia confirmed by chest X-ray or CT scan.
3. RT-PCR Confirmed infection with COVID-19 or strongly suspected infection with pending confirmation studies.
4. Presence of acute respiratory distress syndrome (ARDS).
5. Having either peripheral capillary oxygen saturation (SpO2) ≤ 94% ambient air, or a partial oxygen pressure (PaO2) to fraction of inspired oxygen (FiO2) ratio ≤ 300 mmHg.

Exclusion Criteria:

1. Vitamin D supplementation in the previous month.
2. Contraindication for vitamin D supplementation: active granulomatosis (sarcoidosis, tuberculosis, lymphoma), history of calcic lithiasis, known hypervitaminosis D or hypercalcemia, known intolerance to vitamin D.
3. Organ failure requiring admission to a resuscitation or high dependency unit.
4. Pregnant women.
5. Participation in another simultaneous clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients received the same background treatment for 5 days, following an Institutional protocol for standard of care: hydroxychloroquine 400 mg daily, lopinavir/ritonavir 400/100 mg twice daily or/and remdisivir 200 mg LD then 100 once daily as a maintenance dose and anti-coagulation prophylaxis with enoxaparin subcutaneously once a day if D-dimmer between 500-1000 or enoxaparin therapeutic subcutaneously twice daily if D-dimmer >1000.
Sampling Method: Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Duration of hospitalization | Two weeks
  Length of hospital stay
In-hospital mortality | Two weeks
  Death during hospitalization
Clinical status improvement using six category ordinal scale | Two weeks
  Change in six category ordinal scale. The categories were defined as follows: 1) patient discharged, 2) hospitalization not requiring supplemental oxygen, 3) hospitalization requiring supplemental low-flow oxygen, 4) hospitalization requiring high-flow supplemental oxygen, 5) hospitalization requiring invasive mechanical ventilation, 6) death.
Change in gas exchange | Two weeks
  Difference between ratio of partial pressure of arterial oxygen (PaO2) to the fraction of inspired oxygen (FiO2) at baseline, and before discharge
Time to increase in oxygenation | 48 hours
  Time to increase in SpO2/FiO2 of 50 or greater compared to the baseline SpO2/FiO2)

SECONDARY OUTCOMES:
Change in Lactate dehydrogenase (LDH) levels | Two weeks
  Change in levels of Lactate dehydrogenase (LDH) between baseline and before discharge
Change in C-reactive protein (CRP) levels | Two weeks
  Change in levels of C-reactive protein (CRP) between baseline and before discharge
Change in serum ferritin levels | Two weeks
  Change in levels of serum ferritin between baseline and before discharge
Occurrence of secondary infection | Two weeks
  Occurrence of sepsis
Occurrence of at least one severe adverse event | Two weeks
  Any serious or severe adverse event that might happens during hospital stay
Need for mechanical ventilator or intensive care unit (ICU) support | Two weeks
  Admission to ICU or usage of mechanical ventilator

CONTACTS AND LOCATIONS:
Overall Officials: Neven Sarhan, PhD, Principal Investigator — Misr International University
Locations (1):
- Teachers Hospital, Cairo, Please Select, Egypt

IPD SHARING:
Plan to Share IPD: No